CLINICAL TRIAL: NCT00631358
Title: Assessment of Inflammatory Biomarkers Expressed in a Sjogren's Population: Effect of a Topical Steroid Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Ravaughn Williams, OD, MS, Alcon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORE 14351; NCT00806702 (obsolete NCT alias)
Record Dates: First submitted 2008-02-29; First posted 2008-03-07 (Estimated); Results first posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-03

CONDITIONS: Sjogren's Syndrome
Keywords: Ocular inflammation
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maxidex (Experimental): Maxidex
  Interventions: Drug: Maxidex
- No treatment (Sham Comparator): Healthy normal control group receiving no treatment
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Maxidex — Maxidex (0.1% Dexamethasone) 1 drop in each eye 2 times daily
  Arms: Maxidex
Other: No treatment — Healthy normal control group receiving no treatment
  Arms: No treatment

SUMMARY:
The primary purpose of this study is to quantify the change in expression of biomarkers on the ocular surface of Sjogren's Syndrome participants after treatment with Maxidex.

ELIGIBILITY:
Inclusion Criteria of Sjorgren's Population:

Inclusion Criteria:

* 17 years or older
* LogMar visual acuity of 0.6 or better
* Ocular inflammation associated with Sjogren's Syndrome

Exclusion Criteria:

* Has had an adverse reaction to either topical of systemic steroids in the past
* Has diabetes (type 1 or 2)
* Has glaucoma or evidence of ocular hypertension in either eye or treatment of either within six months of Visit 1
* Has worn contact lenses within one week prior to Visit 1
* Has received ocular prescription therapy in the last 30 days
* Has active ocular infections or inflammation not associated with Sjogren's Syndrome.
* Has any finding in the vitreous, macula, retina or choroid that show signs of inflammation and/or any structural change that in the opinion of the investigator is considered abnormal or unstable for that participant

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Toronto, Toronto
  - Waterloo, Waterloo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited via flyers, newspaper advertisements, radio advertisements and chart review in the doctors' office.
Groups:
- Maxidex: Maxidex 1 drop in each eye 2 times daily
Period: Overall Study
Arm/Group | Maxidex | No Treatment
Started | 50 | 47
Completed | 44 | 45
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maxidex | No Treatment | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 41 | 76
  >=65 years | 15 | 6 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 91
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of Biomarkers After Dosing With Maxidex
Description: Biomarkers are an indicatior of inflammation. In this study, the level of biomarkers before and after anti-inflammatory treatment (Maxidex) is measured for the treatment group. In the control group, the biomarker level is measured at baseline and 2 weeks later. ddCt (Delta-Delta-Ct) is the number of polymerase chain reaction (PCR) cycles required to generate a quantifiable number.
Time Frame: Baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: ddCt (Delta-Delta-Ct)
Arm/Group | Maxidex | No Treatment
Number analyzed (Participants) | 50 | 47
ddCt (Delta-Delta-Ct)
  Baseline | -1.244 (1.08) | -0.29 (0.88)
  2 weeks | -0.033 (1.06) | -0.33 (0.85)

2. Secondary Outcome: Correlation Between Biomarker Expression and Ocular Symptoms
Description: Correlation factor: tumor necrosis factor (TNF) messenger RNA (mRNA) vs. OSDI (Ocular Surface Disease Index).
Time Frame: Baseline to 2 weeks
Measure: Number; unit: Correlation factor
Arm/Group | Maxidex | No Treatment
Number analyzed (Participants) | 50 | 47
Correlation factor | -0.09 | -0.10

3. Secondary Outcome: Correlation Between Biomarker Expression and Tear Film Break up Time
Description: Correlation factor:
  TNFmRNA vs. TFBUT (Tear Film Break-up Time)
Time Frame: Baseline to 2 weeks
Measure: Number; unit: Correlation factor
Arm/Group | Maxidex | No Treatment
Number analyzed (Participants) | 50 | 47
Correlation factor | -0.16 | 0.12

4. Secondary Outcome: Correlation Between Biomarker Expression and NaFl (Sodium Fluorescein) Staining
Description: Correlation factor:
  TNFmRNA vs. NaFl staining
Time Frame: Baseline to 2 weeks
Population: No data available for the no treatment group.
Measure: Number; unit: Correlation factor
Arm/Group | Maxidex | No Treatment
Number analyzed (Participants) | 50 | 0
Correlation factor | -0.05 |

5. Secondary Outcome: Correlation Between Biomarker Expression and the Schirmer Test
Description: Correlation factor: TNFmRNA vs. Schirmer
Time Frame: Baseline to 2 weeks
Measure: Number; unit: Correlation Factor
Arm/Group | Maxidex | No Treatment
Number analyzed (Participants) | 50 | 47
Correlation Factor | -0.02 | 0.07

ADVERSE EVENTS:
Time Frame: Adverse reporting began once the patient enrolled into the study and went on for the duration of the study (6 weeks).
Arm/Group | Maxidex | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall be furnished with copies of any proposed disclosure as follows: Published abstracts will be submitted to the sponsor one month prior to submission allowing the sponsor three weeks to respond. Presentations will be submitted to the sponsor one moth prior to submission allowing the sponsor three weeks to respond. Publications will be submitted to the sponsor two months prior to submission allowing the sponsor two months to respond.